CLINICAL TRIAL: NCT01893060
Title: Umbilical Cord Care for the Prevention of Colonization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, David A Kaufman, Medical Doctor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16859
Record Dates: First submitted 2013-06-20; First posted 2013-07-08 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Line Insertion Site; Central Line-associated Bloodstream Infection (CLABSI)
Keywords: Prematurity; Central line care; Umbilical line colonization; Colonization; Newborn Intensive Care Unit; Neonatal Intensive Care Unit
MeSH Terms: conditions — Premature Birth | interventions — Povidone-Iodine; chlorhexidine gluconate; Poloxamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Povidone-Iodine (Experimental): Umbilical stump care. Povidone-Iodine, USP, Swabstick Singles, applied twice a day to cord stump while umbilical line(s) are in place
  Interventions: Drug: Povidone-Iodine
- Chlorhexidine (Experimental): Umbilical stump care. ChloraPrep® Chlorhexidine Gluconate 2% w/v; 70% Isopropyl Alcohol v/v Swabstick Single, applied twice a day to cord stump while umbilical line(s) are in place
  Interventions: Drug: Chlorhexidine gluconate
- Pluronic Cream (Experimental): Umbilical stump care. Pluronic gel - (F68, Polymyxin, Nystatin, Nitrofurantoin), applied twice a day to cord stump while umbilical line(s) are in place
  Interventions: Drug: Pluronic Cream
- Control (Sham Comparator): No product is applied to cord stump while umbilical line(s) are in place. This is the current standard of care at UVA.
  Interventions: Other: control

INTERVENTIONS:
Drug: Povidone-Iodine — Povidone-Iodine, USP, Swabstick Singles, applied twice a day to cord stump while umbilical line(s) are in place
  Other Names: Betadine
  Arms: Povidone-Iodine
Drug: Chlorhexidine gluconate — Chlorhexidine Gluconate 2% w/v; 70% Isopropyl Alcohol v/v Swabstick Single, applied twice a day to cord stump while umbilical line(s) are in place
  Other Names: ChloraPrep®
  Arms: Chlorhexidine
Drug: Pluronic Cream — Pluronic cream - (F68, Polymyxin, Nystatin, Nitrofurantoin )applied twice a day to cord stump while umbilical line(s) are in place
  Other Names: Pluronic Gel; Pluronic
  Arms: Pluronic Cream
Other: control — No product is applied to cord stump while umbilical line(s) are in place. This is the current standard of care at UVA.
  Other Names: Sham control
  Arms: Control

SUMMARY:
Umbilical catheters are necessary for many infants admitted to the Newborn Intensive Care Unit (NICU)and utilized when indicated for up to 7 to 14 days. Bacterial colonization can occur at the umbilical stump and potentially lead to serious bloodstream infections (BSIs). This study is a prospective, randomized controlled feasibility trial to evaluate three types of hygiene products on umbilical line stumps, on the effect of line colonization and subsequent infections. Infants admitted to the NICU with an umbilical line(s) will be randomized into one of four study groups, three products against standard of care (no product). The three products that will be evaluated are currently being used in different capacities for skin care in the University of Virginia (UVA) NICU. The study hypothesizes that twice daily topical application of 1 or more antiseptic to the top of the umbilical stump will decrease colonization of the umbilical stump while umbilical lines are in place.

DETAILED DESCRIPTION:
Umbilical catheter associated infections are higher (4.4 vs. 3.4 CLABSIs per 1000 line days) than other central lines such as peripherally inserted central catheters (PICCs) and surgically placed central venous lines (CVL) in the NICU. (www.CDC.gov - NSHN 2010 Report). Routine care of the skin entry site (e.g. central line dressing care) is standard for other central lines, but there is no standard for care of the umbilical stump while umbilical lines are in place.

In a pilot study to evaluate the relationship of umbilical stump colonization with gestational age, the number of days the catheter was in place, and the type of organisms, colonization was detected in 78% of patients. There was a direct correlation with colonization and line days as well as an inverse relationship with lower gestational age.

This pilot data supported the need for the study of interventions to reduce umbilical stump colonization, which may help decrease blood stream infections (BSIs) associated with umbilical lines in the NICU. The proposed study will evaluate feasibility of twice daily product application.

ELIGIBILITY:
Inclusion Criteria:

*≤7 days of life

*Umbilical line(s) in place (Umbilical arterial catheter=UAC and/or Umbilical venous catheter=UVC)

Exclusion Criteria:

*Not meeting inclusion criteria

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Colonization of umbilical stump | While umbilical lines are in place, average of 7 days

SECONDARY OUTCOMES:
Late-onset infection | up to 120 days of life, transfer, death or discharge from NICU
  Late-onset infections include BSI, urinary tract infection (UTI), and meningitis. Catheter associated blood stream infections (CLABSI) for this study will be defined as growth in 1 or more blood cultures of any organism including CONS during or within 48-72 hours of having a central line in place, with signs and symptoms of sepsis, and treated for 7 days. Additionally we will compare the CDC definition of CLABSI between groups, and length of stay (LOS).
Contact dermatitis of cord or skin base | while lines are in place, average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: David A Kaufman, MD, Principal Investigator — UVA School of Medicine
Locations (1):
- University of Virginia HealthSystem, Charlottesville, Virginia, United States